CLINICAL TRIAL: NCT00097942
Title: A Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Memantine as Adjunctive Treatment to Atypical Antipsychotics in Schizophrenia Patients With Persistent Residual Symptoms
Brief Title: Evaluation of the Safety and Efficacy of Memantine as Adjunctive Treatment in Schizophrenia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEM-MD-29
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia
Keywords: memantine; adjunctive therapy; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Memantine

INTERVENTIONS:
Drug: memantine HCl

SUMMARY:
Standard antipsychotic drug regimens do not fully address the impact of cognitive symptoms associated with schizophrenia. The NMDA receptor has been connected to the pathophysiology of schizophrenia. Memantine is an uncompetitive NMDA receptor antagonist. It is hypothesized that adjunctive therapy with memantine will reduce NMDA receptor hyperactivity, improving signal to noise ratio and thereby improving cognitive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosed Schizophrenia or schizoaffective disorder who are on a stable antipsychotic regimen with Brief Psychiatric Rating Scale (BPRS) total score greater than or equal to 26 and greater than or equal to 4 on at least one item

Exclusion Criteria:

* Secondary diagnosis of Bipolar I disorder
* Suicidal history
* Organic brain disease
* Dementia
* History of substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2004-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS) - Total Score

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S)
PANNS - Positive Score
PANSS - Negative Score
Calgary Depression Scale for Schizophrenia
Brief Assessment of Cognition
Clinical Global Impression - Improvement

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Synergy Clinical Research, National City, California
  - VA San Diego Healthcare System, San Diego, California
  - University of Miami Jackson Memorial Hospital, Miami, Florida
  - University of Iowa Psychiatric Research, Iowa City, Iowa
  - CBH Health, LLC, Rockville, Maryland
  - Metropolitan Psychiatric Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical School, Lebanon, New Hampshire
  - Nathan Kline Institute, Orangeburg, New York
  - Duke University John Umstead Hospital, Butner, North Carolina
  - UNC - Chapel Hill, Clinical Research Unit, Raleigh, North Carolina
  - University of Cincinnati Medical Science Building, Cincinnati, Ohio
  - University Hills Clinical Research, Irving, Texas
  - Medication Research Clinic, San Antonio, Texas